CLINICAL TRIAL: NCT06198660
Title: Positional Release Technique Versus Cognitive Behavioral Therapy on Chronic Non Specific Low Back Pain
Brief Title: PRT Versus CBT on Chronic Non Specific LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nosaiba Ahmed fahmy Eissa, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRT V CBT IN CNLBP
Record Dates: First submitted 2023-12-18; First posted 2024-01-10 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Chronic Non Specific Mechanical Low Back Pain
Keywords: positional release; cognitive behavioral therapy
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- positional release (Experimental): positional release techniques in addition to conventional physical therapy
  Interventions: Other: positional release technique
- cognitive behavioral therapy (Experimental): cognitive behavioral therapy in addition to conventional physical therapy
  Interventions: Other: cognitive behavioral therapy
- conventional physical therapy (Active Comparator): conventional physical therapy in control group
  Interventions: Other: positional release technique; Other: cognitive behavioral therapy; Other: conventional therapy only

INTERVENTIONS:
Other: positional release technique — positional release techniques in addition to conventional therapy two sessions per week for 6 weeks
  Arms: conventional physical therapy; positional release
Other: cognitive behavioral therapy — cognitive behavioral therapy in addition to conventional therapy two sessions per week for 6 weeks
  Arms: cognitive behavioral therapy; conventional physical therapy
Other: conventional therapy only — conventional therapy two sessions for 6 weeks
  Arms: conventional physical therapy

SUMMARY:
The goal of this clinical trial is to compare between the effect of positional release technique and cognitive behavioral therapy in patients with chronic non specific low back pain.

The main question aims to answer :Is there any differences of using positional release techniques versus cognitive behavioral therapy on patients with chronic low back pain?

DETAILED DESCRIPTION:
Design of the study :

Pretest-posttest randomized controlled trial.

Subjects selection :

sixty patients their age between 25-45 years of both genders with chronic non specific low back pain will participate in this study according tosample size calculation.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be clinically diagnosed with chronic non specific low back pain .
* Their ages will range from 20to40years old.
* body mass index will range from 18 to 30 kg/cm².
* Cognitive score will be 23 or above .
* Voluntary acceptance of participation in this study.

Exclusion Criteria:

* Lumbar canal stenosis
* Lumbar discogenic lesions
* Lumbar infections,tumors.arthiritis
* Patients with decreased range of motion due to congenital anamolies.
* Cognitive and emotional disturbances

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
pressure algometer | pre intervention and immediately after intervention
  change in pain pressure threshold .with unit of measurement kg/cm2

SECONDARY OUTCOMES:
the arabic version of oswestry disability questionnaire | pre intervention and immediately after intervention
  the patients choose one out of six senteces 10 multiple choise questions for back pain higher scores indicate great pain

CONTACTS AND LOCATIONS:
Overall Officials: Nosaiba Eissa, Principal Investigator — Cairo University
Locations (1):
- Horus University, Damietta, New Damietta, Egypt